CLINICAL TRIAL: NCT03301948
Title: The Effects of a Single Day of Mixed Macronutrient Overfeeding on Energy Balance and Metabolic Responses in Healthy Young Men
Brief Title: Effects of a Single Day of Mixed Macronutrient Overfeeding on Energy Balance and Metabolic Responses
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Leeds Beckett University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Prevention
Other Study IDs: 34693
Record Dates: First submitted 2017-08-08; First posted 2017-10-04 (Actual); Last update posted 2019-01-14 (Actual); Status verified 2019-01

CONDITIONS: Metabolic Disease; Appetitive Behavior
MeSH Terms: conditions — Metabolic Diseases; Appetitive Behavior

STUDY DESIGN:
Intervention Model Description: Single blind, counterbalanced, crossover trial
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Overfeed (Experimental): Experimental trial where participants are provided with 50% higher energy intake than their estimated requirements on the first day of the trial.
  Interventions: Other: Overfeed
- Energy Balance (Experimental): Experimental trial where participants are provided with an energy intake equal to their estimated requirements on the first day of the trial.
  Interventions: Other: Energy Balance

INTERVENTIONS:
Other: Overfeed — Participants consume energy intakes that are 50% higher than their estimated requirements instead of consuming energy intakes equal to their estimated requirements
  Arms: Overfeed
Other: Energy Balance — Participants consume energy intakes equal to their estimated requirements instead of consuming intakes that are 50% higher than their estimated requirements
  Arms: Energy Balance

SUMMARY:
Healthy male participants are recruited to observe potentially deleterious changes in appetite regulation and metabolic control. Participants will be provided with an energy intake representative of their daily requirements on the first day of one trial and will be provided with an additional 50% energy intake on the first day of another trial. Outcome variables will be assessed during the second day of each trial in response to a fixed mixed macronutrient meal tolerance test.

DETAILED DESCRIPTION:
All testing will take place within the Carnegie Research Institute, Leeds Beckett University. We will ask all the participants to visit on five occasions for the completion of a preliminary screening trial and two single-blind counterbalanced experimental trials which each require the participants to visit the laboratory on two consecutive days. The experimental trials will be separated by a minimum of one week.

Visit 1: Preliminary Screening:

Before an individual can take part in the experiment, they will need to undergo screening. Individuals will need to complete a Health Screen Questionnaire. Individuals will be excluded from the study if they are not currently in good health, have any condition that would alter their metabolism and/or have had significant medical problems in the past that may affect the outcomes of the study. Individuals will also be asked to be complete a Three-Factor Eating Questionnaire, to check that they are not restrained eaters, and an International Physical Activity Questionnaire (IPAQ) to ensure that all participants are either sedentary or moderately active. All individuals will be asked to confirm that they have been weight stable for at least six months before participating and that they are not currently dieting. Height, body mass and age will be collected to calculate the energy requirements for the main trials based on the Mifflin equation.

Visits 2, 3, 4 and 5: Experimental Trials:

The participants will be asked to record their food intakes and activity patterns during the three days prior to the first experimental test using a food and physical activity diary. They will then be instructed to repeat this diet and activity pattern prior to the second experimental trial. Participants will be required to arrive at the laboratory for all experimental trials after an overnight fast of at least 10 hours and having refrained from any strenuous activity for 48 hours, and alcohol and caffeine consumption in the previous 24 hours. Two hours before arriving at the laboratory on the day of the experimental trials, participants will be required to ingest 300 mL of water to standardise hydration levels for the trial.

During Day One of each experimental trial, participants will consume a porridge-based breakfast, soup- and pasta-based lunch, and rice-based evening meal under laboratory observation. The meals will contain macronutrient contents representative of current dietary recommendations of 50% carbohydrate, 15% protein and 35% fat. These meals have been selected to facilitate manipulation of the energy content, while matching the meals for appearance and palatability. During one trial, these meals will provide the calculated energy requirement for each individual based on the Mifflin equation and a physical activity factor of 1.4. The meals will be covertly manipulated to provide an additional 50% energy intake during the other trial. The provision of 150% of the estimated energy requirements for participants has been used in previous research for five day periods but will only be provided for a single day in the present study. Participants will be required to consume all of the diet during the standardised phase (i.e. either their daily energy requirements or the 50% overfeed) and will be blinded to the energy content of the trials. After the consumption of the evening meal (~6pm), participants will have fulfilled the requirements for day one and will be asked not to consume any food prior to returning to the laboratory between 7am and 9am the next morning.

On Day Two of each experimental trial day, participants will arrive at the laboratory after an overnight fast and an Introcan Safety Cannula will be placed into a vein in the anticubital space for regular venous blood sampling. Blood samples will be collected in the fasted state and every 30 min after consumption of a standardised breakfast for a period of three hours. After the collection of the final blood sample, the cannula will be removed and participants will be provided with an ad libitum pasta meal (50% carbohydrate, 15% protein, 35% fat) for the assessment of energy intake. Participants will consume ad libitum meals in isolation to prevent any social influences and will be instructed to eat until 'satisfied'.

ELIGIBILITY:
Inclusion Criteria:

* weight stable
* healthy

Exclusion Criteria:

* any personal history of cardiovascular or metabolic disease
* smokers
* currently dieting
* taking any medication known to influence appetite or metabolic outcomes
* highly active (IPAQ category 3)

Ages: 18 Years to 35 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 12 (Actual)
Dates: Start 2017-05-01 (Actual); Primary Completion 2019-01-11 (Actual); Study Completion 2019-01-11 (Actual)

PRIMARY OUTCOMES:
Appetite perceptions assessed using 100mm visual analogue scales | 28 hours
  Appetite perceptions using 100mm visual analogue scales
Ad libitum energy intake | 28 hours
  Ad libitum energy intake using an ad libitum pasta meal
Plasma acylated ghrelin concentrations | 28 hours
  Measured using ELISA from venous blood samples
Plasma peptide YY concentrations | 28 hours
  Measured using ELISA from venous blood samples
Plasma GLP-1 concentrations | 28 hours
  Measured using ELISA from venous blood samples

SECONDARY OUTCOMES:
Palatability perceptions assessed using 100mm visual analogue scales | 28 hours
  Palatability of the test meals assessed via 100mm visual analogue scales during the first day of each trial
Blinding assessment | One week
  To assess whether the blinding of dietary manipulation of the first day of each trial was successful. This will be assessed via an exit questionnaire which requires qualitative responses regarding any noticeable differences in the foods provided and what aspect of the food the participants thought had been manipulated during the trials.
Plasma insulin concentrations | 28 hours
  Measured using ELISA from venous blood samples
Plasma glucose concentrations | 28 hours
  Measured using photometric analysis from venous blood samples
Plasma triglyceride concentrations | 28 hours
  Measured using photometric analysis from venous blood samples

CONTACTS AND LOCATIONS:
Overall Officials: Kevin Deighton, PhD, Principal Investigator — Leeds Beckett University
Locations (1):
- Leeds Beckett University, Leeds, United Kingdom

IPD SHARING:
Plan to Share IPD: No